CLINICAL TRIAL: NCT04414943
Title: Effects of Low-dose S-ketamine on the Incidence of Postpartum Depression in Women With Prenatal Depression: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Low-dose S-ketamine in Women With Prenatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University International Hospital (Other); Hunan Provincial Maternal and Child Health Care Hospital (Other); Nanjing Medical University (Other); Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019[336]
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Prenatal Depression; Ketamine; Postpartum Depression
Keywords: Prenatal Depression; S-ketamine; Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-katamine group (Experimental): For women in this group, study drug (s-ketamine 0.2 mg/kg in 20 ml normal saline) will be infused at a rate of 30 ml/h (infusion finished in 40 minutes) after giving birth. Women will be monitored for 60 minutes and then sent back to the ward.
  Interventions: Drug: S-ketamine
- Placebo group (Placebo Comparator): For women in this group, study drug (20 ml normal saline) will be infused at a rate of 30 ml/h (infusion finished in 40 minutes) after giving birth. Women will be monitored for 60 minutes and then sent back to the ward.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-ketamine — For women in this group, active drug (s-ketamine 0.2 mg/kg in 20 ml normal saline) will be infused at a rate of 30 ml/h (infusion finished in 40 minutes) after giving birth. They will be monitored for 60 minutes and then sent back to the ward.
  Other Names: S-ketamine hydrochloride
  Arms: S-katamine group
Drug: Placebo — For women in this group, placebo (20 ml normal saline) will be infused at a rate of 30 ml/h (infusion finished in 40 minutes) after giving birth. They will be monitored for 60 minutes and then sent back to the ward.
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
Prenatal depression is an important risk factor of postpartum depression. Low-dose ketamine has been used for depression treatment. As a stereoisomer of ketamine, s-ketamine has similar effects to ketamine in anti-depression. We speculate that, for pregnant women with prenatal depression, low-dose s-ketamine infusion after childbirth may reduce the incidence of postpartum depression.

DETAILED DESCRIPTION:
Studies have shown that prenatal depression symptoms are important predictors of postpartum depression. Screening of pregnant women's mental condition before giving birth, early identification of pregnant women with symptoms of prenatal depression, and providing appropriate interventions may play an important role in reducing the incidence of postpartum depression. Ketamine is an NMDA-receptor antagonist. In recent years, many studies confirmed that ketamine has a significant antidepressant effect. As a stereoisomer of ketamine, s-ketamine has similar effects to ketamine in anti-depression. In clinical application, s-ketamine has stronger analgesic effect, better anesthetic effect and lower incidence of adverse psychological reactions. We speculate that, for pregnant women with prenatal depression, low-dose s-ketamine infusions after childbirth may reduce postpartum depression. Evidence is lacking in this regard.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age ≥18 years;
2. Prenatal Edinburgh postnatal depression scale score ≥10 points.

Exclusion Criteria:

1. A clear history of mental illness (depression, schizophrenia, etc.) or communication difficulties;
2. Severe pregnancy complications, such as severe preeclampsia, placental implantation, HELLP (syndrome hemolytic anemia, elevated liver function and low platelet count) syndrom, placenta previa, and placental abruption;
3. American Society of Anesthesiologists classification ≥III;
4. Presence of contraindications to ketamine/s-ketamine use, such as refractory hypertension, severe cardiovascular disease (New York Heart Association classification ≥III), and hyperthyroidism.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This clinical trail is based in pregnant women.
Enrollment: 364 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
The incidence of depression at 42 days postpartum. | At 42 days after childbirth.
  Depression at 42 days postpartum will be diagnosed by psychiatrists according to the Mini-International Neuropsychiatric Interview (MINI)-6.0.

SECONDARY OUTCOMES:
Maternal depression score at 7 days postpartum. | At 7 days after childbirth.
  Maternal depression will be assessed with the Edinburgh Postnatal Depression Scale (EPDS; score range 0-30, with higher score indicating more severe depression). The assessment will be conducted by a telephone interview.
Maternal depression score at 42 days postpartum. | At 42 days after childbirth.
  Maternal depression will be assessed with the Edinburgh Postnatal Depression Scale (EPDS; score range 0-30, with higher score indicating more severe depression). The assessment will be conducted by a face-to-face interview or an online video interview.
Maternal depression severity at 42 days postpartum. | At 42 days after childbirth.
  Maternal depression severity will be assessed with the Hamilton Depression Scale-17 (HAMD; score range 0-52, with higher score indicating more severe depression). The assessment will be conducted by a face-to-face interview or an online video interview.
Intensity of pain at 1, 7, and 42 days postpartum. | At 1, 7, and 42 days after childbirth.
  Intensity of pain will be assessed with the numeric rating scale (a 11-point scale where 0=no pain and 10=the worst pain).
Maternal breast feeding at 1, 7, and 42 days postpartum. | At 1, 7, and 42 days after childbirth.
  The mode of baby feeding include breast feeding, mixed feeding, or formula feeding.
Length of hospital stay after giving birth. | Up to 30 days after giving birth.
  Length of hospital stay after giving birth.
Incidence of maternal complications within 42 days postpartum. | Up to 42 days after giving birth.
  Maternal complications are defined as those that are harmful to maternal health and require medical intervention.
Incidence of neonatal diseases within 42 days. | Up to 42 days after birth.
  Neonatal diseases are defined as those that require medical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (7):
- China (7):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - Huaian Maternal and Child Health Care Hospital, Huaian, Jiangsu
  - Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
IPD will be available by contacting Dr. Dong-Xin Wang (wangdongxin@hotmail.com) after the trial is completed.

REFERENCES:
- [Background] Nonacs R, Cohen LS. Postpartum mood disorders: diagnosis and treatment guidelines. J Clin Psychiatry. 1998;59 Suppl 2:34-40. PMID 9559758
- [Background] Kim S, Soeken TA, Cromer SJ, Martinez SR, Hardy LR, Strathearn L. Oxytocin and postpartum depression: delivering on what's known and what's not. Brain Res. 2014 Sep 11;1580:219-32. doi: 10.1016/j.brainres.2013.11.009. Epub 2013 Nov 14. PMID 24239932
- [Background] Giallo R, Pilkington P, McDonald E, Gartland D, Woolhouse H, Brown S. Physical, sexual and social health factors associated with the trajectories of maternal depressive symptoms from pregnancy to 4 years postpartum. Soc Psychiatry Psychiatr Epidemiol. 2017 Jul;52(7):815-828. doi: 10.1007/s00127-017-1387-8. Epub 2017 Apr 27. PMID 28451700
- [Background] Giallo R, Cooklin A, Nicholson JM. Risk factors associated with trajectories of mothers' depressive symptoms across the early parenting period: an Australian population-based longitudinal study. Arch Womens Ment Health. 2014 Apr;17(2):115-25. doi: 10.1007/s00737-014-0411-1. Epub 2014 Jan 15. PMID 24424796
- [Background] Sutter-Dallay AL, Cosnefroy O, Glatigny-Dallay E, Verdoux H, Rascle N. Evolution of perinatal depressive symptoms from pregnancy to two years postpartum in a low-risk sample: the MATQUID cohort. J Affect Disord. 2012 Jun;139(1):23-9. doi: 10.1016/j.jad.2011.08.018. Epub 2012 Mar 11. PMID 22410506
- [Background] McCall-Hosenfeld JS, Phiri K, Schaefer E, Zhu J, Kjerulff K. Trajectories of Depressive Symptoms Throughout the Peri- and Postpartum Period: Results from the First Baby Study. J Womens Health (Larchmt). 2016 Nov;25(11):1112-1121. doi: 10.1089/jwh.2015.5310. Epub 2016 Jun 16. PMID 27310295
- [Background] Tsai R, Schaffir J. Effect of depot medroxyprogesterone acetate on postpartum depression. Contraception. 2010 Aug;82(2):174-7. doi: 10.1016/j.contraception.2010.03.004. Epub 2010 Apr 13. PMID 20654759
- [Background] Ding T, Wang DX, Qu Y, Chen Q, Zhu SN. Epidural labor analgesia is associated with a decreased risk of postpartum depression: a prospective cohort study. Anesth Analg. 2014 Aug;119(2):383-392. doi: 10.1213/ANE.0000000000000107. PMID 24797120
- [Background] Quevedo LA, Silva RA, Godoy R, Jansen K, Matos MB, Tavares Pinheiro KA, Pinheiro RT. The impact of maternal post-partum depression on the language development of children at 12 months. Child Care Health Dev. 2012 May;38(3):420-4. doi: 10.1111/j.1365-2214.2011.01251.x. Epub 2011 Jun 8. PMID 21651606
- [Background] Parsons CE, Young KS, Rochat TJ, Kringelbach ML, Stein A. Postnatal depression and its effects on child development: a review of evidence from low- and middle-income countries. Br Med Bull. 2012;101:57-79. doi: 10.1093/bmb/ldr047. Epub 2011 Nov 29. PMID 22130907
- [Background] Weitzman M, Rosenthal DG, Liu YH. Paternal depressive symptoms and child behavioral or emotional problems in the United States. Pediatrics. 2011 Dec;128(6):1126-34. doi: 10.1542/peds.2010-3034. Epub 2011 Nov 7. PMID 22065273
- [Background] Demontigny F, Girard ME, Lacharite C, Dubeau D, Devault A. Psychosocial factors associated with paternal postnatal depression. J Affect Disord. 2013 Aug 15;150(1):44-9. doi: 10.1016/j.jad.2013.01.048. Epub 2013 Mar 13. PMID 23489392
- [Background] Dietz LJ, Jennings KD, Kelley SA, Marshal M. Maternal depression, paternal psychopathology, and toddlers' behavior problems. J Clin Child Adolesc Psychol. 2009 Jan;38(1):48-61. doi: 10.1080/15374410802575362. PMID 19130357
- [Background] Pawlby S, Sharp D, Hay D, O'Keane V. Postnatal depression and child outcome at 11 years: the importance of accurate diagnosis. J Affect Disord. 2008 Apr;107(1-3):241-5. doi: 10.1016/j.jad.2007.08.002. Epub 2007 Sep 12. PMID 17854906
- [Background] Robertson E, Grace S, Wallington T, Stewart DE. Antenatal risk factors for postpartum depression: a synthesis of recent literature. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):289-95. doi: 10.1016/j.genhosppsych.2004.02.006. PMID 15234824
- [Background] Klainin P, Arthur DG. Postpartum depression in Asian cultures: a literature review. Int J Nurs Stud. 2009 Oct;46(10):1355-73. doi: 10.1016/j.ijnurstu.2009.02.012. Epub 2009 Mar 26. PMID 19327773
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Lee DT, Yip AS, Leung TY, Chung TK. Identifying women at risk of postnatal depression: prospective longitudinal study. Hong Kong Med J. 2000 Dec;6(4):349-54. PMID 11177155
- [Background] Milgrom J, Gemmill AW, Bilszta JL, Hayes B, Barnett B, Brooks J, Ericksen J, Ellwood D, Buist A. Antenatal risk factors for postnatal depression: a large prospective study. J Affect Disord. 2008 May;108(1-2):147-57. doi: 10.1016/j.jad.2007.10.014. Epub 2007 Dec 18. PMID 18067974
- [Background] Siu BW, Leung SS, Ip P, Hung SF, O'Hara MW. Antenatal risk factors for postnatal depression: a prospective study of Chinese women at maternal and child health centres. BMC Psychiatry. 2012 Mar 22;12:22. doi: 10.1186/1471-244X-12-22. PMID 22436053
- [Background] Huynh NN, McIntyre RS. What Are the Implications of the STAR*D Trial for Primary Care? A Review and Synthesis. Prim Care Companion J Clin Psychiatry. 2008;10(2):91-6. doi: 10.4088/pcc.v10n0201. PMID 18458732
- [Background] Schwartz J, Murrough JW, Iosifescu DV. Ketamine for treatment-resistant depression: recent developments and clinical applications. Evid Based Ment Health. 2016 May;19(2):35-8. doi: 10.1136/eb-2016-102355. Epub 2016 Apr 6. PMID 27053196
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Newport DJ, Carpenter LL, McDonald WM, Potash JB, Tohen M, Nemeroff CB; APA Council of Research Task Force on Novel Biomarkers and Treatments. Ketamine and Other NMDA Antagonists: Early Clinical Trials and Possible Mechanisms in Depression. Am J Psychiatry. 2015 Oct;172(10):950-66. doi: 10.1176/appi.ajp.2015.15040465. PMID 26423481
- [Background] Kishimoto T, Chawla JM, Hagi K, Zarate CA, Kane JM, Bauer M, Correll CU. Single-dose infusion ketamine and non-ketamine N-methyl-d-aspartate receptor antagonists for unipolar and bipolar depression: a meta-analysis of efficacy, safety and time trajectories. Psychol Med. 2016 May;46(7):1459-72. doi: 10.1017/S0033291716000064. Epub 2016 Feb 12. PMID 26867988
- [Background] Drewniany E, Han J, Hancock C, Jones RL, Lim J, Nemat Gorgani N, Sperry JK 3rd, Yu HJ, Raffa RB. Rapid-onset antidepressant action of ketamine: potential revolution in understanding and future pharmacologic treatment of depression. J Clin Pharm Ther. 2015 Apr;40(2):125-30. doi: 10.1111/jcpt.12238. Epub 2014 Dec 26. PMID 25545040
- [Background] Strasburger SE, Bhimani PM, Kaabe JH, Krysiak JT, Nanchanatt DL, Nguyen TN, Pough KA, Prince TA, Ramsey NS, Savsani KH, Scandlen L, Cavaretta MJ, Raffa RB. What is the mechanism of Ketamine's rapid-onset antidepressant effect? A concise overview of the surprisingly large number of possibilities. J Clin Pharm Ther. 2017 Apr;42(2):147-154. doi: 10.1111/jcpt.12497. Epub 2017 Jan 22. PMID 28111761
- [Background] Fond G, Loundou A, Rabu C, Macgregor A, Lancon C, Brittner M, Micoulaud-Franchi JA, Richieri R, Courtet P, Abbar M, Roger M, Leboyer M, Boyer L. Ketamine administration in depressive disorders: a systematic review and meta-analysis. Psychopharmacology (Berl). 2014 Sep;231(18):3663-76. doi: 10.1007/s00213-014-3664-5. Epub 2014 Jul 20. PMID 25038867
- [Background] Park M, Niciu MJ, Zarate CA Jr. Novel Glutamatergic Treatments for Severe Mood Disorders. Curr Behav Neurosci Rep. 2015 Dec;2(4):198-208. doi: 10.1007/s40473-015-0050-5. Epub 2015 Oct 9. PMID 26824031
- [Background] Perry EB Jr, Cramer JA, Cho HS, Petrakis IL, Karper LP, Genovese A, O'Donnell E, Krystal JH, D'Souza DC; Yale Ketamine Study Group. Psychiatric safety of ketamine in psychopharmacology research. Psychopharmacology (Berl). 2007 Jun;192(2):253-60. doi: 10.1007/s00213-007-0706-2. Epub 2007 Feb 16. PMID 17458544
- [Background] Xu Y, Li Y, Huang X, Chen D, She B, Ma D. Single bolus low-dose of ketamine does not prevent postpartum depression: a randomized, double-blind, placebo-controlled, prospective clinical trial. Arch Gynecol Obstet. 2017 May;295(5):1167-1174. doi: 10.1007/s00404-017-4334-8. Epub 2017 Mar 29. PMID 28357557
- [Background] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Singh JB, Fedgchin M, Daly E, Xi L, Melman C, De Bruecker G, Tadic A, Sienaert P, Wiegand F, Manji H, Drevets WC, Van Nueten L. Intravenous Esketamine in Adult Treatment-Resistant Depression: A Double-Blind, Double-Randomization, Placebo-Controlled Study. Biol Psychiatry. 2016 Sep 15;80(6):424-431. doi: 10.1016/j.biopsych.2015.10.018. Epub 2015 Nov 3. PMID 26707087
- [Background] Paul R, Schaaff N, Padberg F, Moller HJ, Frodl T. Comparison of racemic ketamine and S-ketamine in treatment-resistant major depression: report of two cases. World J Biol Psychiatry. 2009;10(3):241-4. doi: 10.1080/15622970701714370. PMID 19224412
- [Background] Gaillard A, Le Strat Y, Mandelbrot L, Keita H, Dubertret C. Predictors of postpartum depression: prospective study of 264 women followed during pregnancy and postpartum. Psychiatry Res. 2014 Feb 28;215(2):341-6. doi: 10.1016/j.psychres.2013.10.003. Epub 2013 Nov 6. PMID 24370337
- [Derived] Wang S, Deng CM, Zeng Y, Chen XZ, Li AY, Feng SW, Xu LL, Chen L, Yuan HM, Hu H, Yang T, Han T, Zhang HY, Jiang M, Sun XY, Guo HN, Sessler DI, Wang DX. Efficacy of a single low dose of esketamine after childbirth for mothers with symptoms of prenatal depression: randomised clinical trial. BMJ. 2024 Apr 10;385:e078218. doi: 10.1136/bmj-2023-078218. PMID 38808490